CLINICAL TRIAL: NCT04331990
Title: Efficacy of Adding Mechanical Nonsurgical Knee Traction to Standard Physical Therapy Rehabilitation of Knee Osteoarthritis: a Randomized Controlled Trial
Brief Title: The Distraction of Knee Joint to Alleviate osteoArthritic Pain (DiKAP) Trial
Acronym: DiKAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Prince Sultan Military College of Health Sciences (Other)
Responsible Party: Principal Investigator, Ahmed Farrag, Assistant Professor, Prince Sultan Military College of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PT-2020-02
Record Dates: First submitted 2020-03-29; First posted 2020-04-02 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Knee Osteoarthritis
Keywords: Knee; Osteoarthritis; Pain; Joint distraction
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Both the outcome assessors and the study statistician will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Physical Therapy (Active Comparator): Control group for the study. Intervention in the form of warm-up and strengthening, stretching and neuromuscular control exercises.
  Interventions: Other: Standard Physcial Therapy
- Intermittent Mechanical Traction (Experimental): Standard care in addition to intermittent mechanical distraction of the knee joint.
  Interventions: Other: Intermittent Mechanical Traction
- Continuous Mechanical Traction (Experimental): Standard care in addition to continuous mechanical distraction of the knee joint
  Interventions: Other: Continuous Mechanical Traction

INTERVENTIONS:
Other: Standard Physcial Therapy — Patients assigned to this group will receive a 40-min multimodal supervised physical therapy treatment comprised of warm-up (10-min cycling/walking), muscle strengthening and stretching, and neuromuscular control exercises. Manual mobilization techniques may be applied as necessary according to the findings of the physical examination. Treating physical therapists will prescribe exercises based on a predetermined list of exercises.
  Arms: Standard Physical Therapy
Other: Intermittent Mechanical Traction — In addition to the standard treatment, patients in this group will receive intermittent knee joint decompression for 20 minutes. Patients will be lying supine with the knee semiflexed to 30° and supported by a wedge under the knee. A customized leg cuff will be placed around the lower leg and two ropes will be extending horizontally from the cuff to the vertical traction weight using a pulley system to transfer the traction force to the tibiofemoral articulation. The magnitude of the traction force will be between 10-15% of the patient's body weight. The traction force will be applied for 10 application cycles; each cycle comprised of 2 minutes traction followed by 30 seconds relief. This will sum up to 20 minutes of actual joint traction duration. The traction force application and relief time will be controlled manually by the treating therapist. Knee joint traction procedures will be applied at the end of the physical therapy session.
  Arms: Intermittent Mechanical Traction
Other: Continuous Mechanical Traction — Patients assigned to this group will receive the same treatment protocol as those in the Intermittent Mechanical Traction group. However, the knee traction force will be applied continuously for 20 minutes without intermittent force relief periods.
  Arms: Continuous Mechanical Traction

SUMMARY:
This is a randomized controlled trial examining the short- and long-term effects of mechanical nonsurgical knee joint traction on knee pain, function, and quality of life.

DETAILED DESCRIPTION:
Knee OA symptoms are known to be impacted by increased joint loading and reduced joint space width between the articulating bones.

Objectives:

* Primary objective: Investigate the short- and long-term efficacy of adding nonsurgical knee joint distraction to standard multimodal physical therapy treatment on pain, joint function and quality of life in patients with knee OA compared with standard physical therapy treatment alone.
* Secondary objective: examine whether the efficacy of mechanical traction would differ based on the mode of application (continuous vs. intermittent traction).

Design and Subjects: A prospective, active control, three-parallel-group, investigator-blinded, randomized controlled trial. 198 subjects will be recruited and randomly assigned to one of three study groups at a 1:1:1 allocation ratio (66 participants per group): a) Standard care only, b) continuous mechanical traction plus standard care, and c) intermittent mechanical traction plus standard care.

Intervention: Participants in the standard care only group will receive 16 treatment sessions (2sessions/week) over 8 weeks, followed by 4 booster sessions (1session/2months) during the one-year period of the trial. Mechanical traction groups will receive standard care in addition to 20-minute knee traction (continuous or intermittent) using an external weight applying knee traction force.

Outcome measures: The primary outcomes are physical function and pain assessed using the Knee Injury and Osteoarthritis Outcome Score (KOOS). Secondary outcomes include the Numeric Pain Rating Scale, quality of life, Timed Up and Go, 40m fast-paced walk, and 30s chair stand tests, patient's self-perceived efficacy of treatment and patient's global assessment.

Data Analysis: Data will be analyzed using the intension-to-treat (ITT) analysis with multiple imputations. The per-protocol analysis will be carried out and reported if its findings are different from those of the primary ITT analysis. The primary analysis of the primary outcomes at two- and six-month follow-up time points will be carried out using analysis of covariance (ANCOVA) test with adjustment for a set of pre-specified baseline covariates. Secondary analysis using ANCOVA test for the primary outcomes at the 12-month time point, and secondary outcomes at all follow-up time points will also be carried out.

ELIGIBILITY:
Inclusion Criteria:

* ≥40 years of age;
* having knee pain;
* having at least three of the following additional symptoms: a-morning stiffness ≤ 30 minutes, b-crepitation, c-bone margin tenderness, d-bony enlargement or e-no palpable warmth;
* willing to provide informed consent

Exclusion Criteria:

* rheumatoid arthritis;
* serious pathological conditions (inflammatory arthritis and malignancy); total or partial arthroplasty of the affected knee joint, or on waiting list for joint replacement surgery;
* recent surgical procedure of the lower extremities in the previous 6 months;
* uncontrolled hypertension and unstable cardiovascular problems that could subject the participant to increased risk with exercise and physical exertion;
* physical incapability to safely perform exercises, walking or stationary cycling, as in: debilitating visual defects, neurological problems, exaggerated low back pain, advanced osteoporosis, and inability to walk 10 meters without an assistive device;
* use of prescribed analgesics, corticosteroid or analgesic injection intervention for knee pain within the previous 30 days;
* lack of clear comprehension of study procedures or inability to comply with instructions;
* stated inability to attend or complete the proposed course of intervention and follow-up schedule.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in pain score using the Arabic version of the Knee Injury and Osteoarthritis Outcome Score (KOOS) | Baseline, 2, 6 and 12 months follow-up
  A 5-point Likert scale comprised of 42 questions across 5 subscales. Standardized answers are assigned a score from 0 (no symptoms) to 4 (extreme symptoms). A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Change in physical function score using the Arabic version of the Knee Injury and Osteoarthritis Outcome Score (KOOS) | Baseline, 2, 6 and 12 months follow-up
  A 5-point Likert scale comprised of 42 questions across 5 subscales. Standardized answers are assigned a score from 0 (no symptoms) to 4 (extreme symptoms). A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.

SECONDARY OUTCOMES:
Change in knee pain using the Arabic version of the Numeric Pain Rating Scale (ANPRS) | Baseline, 2, 6 and 12 months follow-up
  A horizontal 11-point scale (0-10), with 0 indicating no pain and 10 indicating the worst pain ever.
Change in Patient's Global Assessment | 2, 6, 12 months follow-up
  A single question using a 7-point Likert scale (1 indicates much worse, and 7 indicates much better).
Change in Health-related Quality of Life score using the Arabic version of the Short Form 36 (SF-36) scale | Baseline, 2, 6 and 12 months follow-up
  A 36-item scale with a score ranging from 0 (worst health status) to 100 (best health status).
Change in the time taken to complete the Timed Up and Go (TUG) | Baseline, 2, 6 and 12 months follow-up
  Time (seconds) taken to rise from a chair, walk 3m, turn, walk back to the chair, then sit down
Change in the wakling speed for the 40m fast-paced walk test | Baseline, 2, 6 and 12 months follow-up
  The walking speed (m/s) will be recorded to walk quickly and safely over a 10m walkway for a total of 40m (4 x 10m).
Change in number of repetitions during the 30s chair stand test | Baseline, 2, 6 and 12 months follow-up
  The maximum number of chair stand repetitions possible in a 30 second period is counted and recorded.
change in the Patient's Self-perceived Efficacy of treatment | 2, 6 and 12 months follow-up
  A single question inquiring about the patient's perception regarding the effectiveness of physical therapy intervention to improve the OA symptoms. A 5-point Likert scale (1 indicates not effective, and 5 indicates greatly effective).
Change in other subscales of the Knee Injury and Osteoarthritis Outcome Score (KOOS (Symptoms, Sport and Recreation Function, and knee-related Quality of Life). | Baseline, 2, 6 and 12 months follow-up
  A 5-point Likert scale comprised of 42 questions across 5 subscales. Standardized answers are assigned a score from 0 (no symptoms) to 4 (extreme symptoms). A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.

OTHER OUTCOMES:
Number of sessions attended by the patient | 2, 6, 12 months follow-up
  Patient adherence to physical therapy sessions will be recorded in the patient's file. Adherence to the home exercise program will be self-reported by the patient in a home exercise logbook.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Farrag, PhD, Principal Investigator — Prince Sultan Military College of Health Sciences

IPD SHARING:
Plan to Share IPD: No